CLINICAL TRIAL: NCT01529645
Title: Phase I, Randomized, Controlled, Observer-Blind, Dose-Ranging Study of Acellular Pertussis and Tetanus-Diptheria-Acellular Pertussis Booster Vaccine in Adults Ages 18 to 40 Years.
Brief Title: Safety and Dose Ranging Study of Acellular Pertussis and Acellular Pertussis -Tetanus-Diphtheria Booster Vaccines in Healthy Adults Ages 18 to 40 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V113_01; 2011-000688-28 (EudraCT Number)
Record Dates: First submitted 2012-02-06; First posted 2012-02-09 (Estimated); Results first posted 2014-09-18 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Pertussis; Whooping Cough; Tetanus; Lockjaw; Diphtheria
Keywords: pertussis; booster vaccine; tetanus; diphtheria in adults
MeSH Terms: conditions — Whooping Cough; Tetanus; Trismus; Diphtheria | interventions — Tetanus Toxoid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (10):
- Group 1: aP booster (Experimental): Subjects received acellular pertussis (aP) vaccine with different antigen dose formulations: low dose of PT, FHA, PRN, followed by one fixed dose of diphtheria and tetanus vaccine (adsorbed, reduced antigen content, Germany) administered one month apart.
  Interventions: Biological: Acellular pertussis vaccine; Biological: Diphtheria and tetanus vaccine (adsorbed, reduced antigen content, Germany)
- Group 2: aP booster (Experimental): Subjects received acellular pertussis (aP) vaccine with different antigen dose formulations: medium dose of PT, FHA, PRN, followed by one fixed dose of diphtheria and tetanus vaccine (adsorbed, reduced antigen content, Germany) administered one month apart.
  Interventions: Biological: Acellular pertussis vaccine; Biological: Diphtheria and tetanus vaccine (adsorbed, reduced antigen content, Germany)
- Group 3: aP booster (Experimental): Subjects received acellular pertussis (aP) vaccine with different antigen dose formulations: high dose of PT, FHA, PRN, followed by one fixed dose of diphtheria and tetanus vaccine (adsorbed, reduced antigen content, Germany) administered one month apart.
  Interventions: Biological: Acellular pertussis vaccine; Biological: Diphtheria and tetanus vaccine (adsorbed, reduced antigen content, Germany)
- Group 4: TdaP booster (Experimental): Subjects received tetanus, reduced diphtheria, and acellular pertussis vaccine (adsorbed) with different antigen dose formulations: low dose of PT, FHA, PRN, low dose of D (diphteria) toxoid, fixed dose of T (tetanus) toxoid, followed by one administration of saline solution one month apart.
  Interventions: Biological: Tetanus, reduced diphtheria, and acellular pertussis vaccine (adsorbed); Other: Saline solution
- Group 5: TdaP booster (Experimental): Subjects received tetanus, reduced diphtheria, and acellular pertussis vaccine (adsorbed) with different antigen dose formulations: medium dose of PT, FHA, PRN, low dose of D toxoid, fixed dose of T toxoid, followed by one administration of saline solution one month apart.
  Interventions: Biological: Tetanus, reduced diphtheria, and acellular pertussis vaccine (adsorbed); Other: Saline solution
- Group 6: TdaP booster (Experimental): Subjects received tetanus, reduced diphtheria, and acellular pertussis vaccine (adsorbed) with different antigen dose formulations: high dose of PT, FHA, PRN, low dose of D toxoid, fixed dose of T toxoid, followed by one administration of saline solution one month apart.
  Interventions: Biological: Tetanus, reduced diphtheria, and acellular pertussis vaccine (adsorbed); Other: Saline solution
- Group 7: TdaP booster (Experimental): Subjects received tetanus, reduced diphtheria, and acellular pertussis vaccine (adsorbed) with different antigen dose formulations: low dose of PT, FHA, PRN, double dose of D toxoid, fixed dose of T toxoid, followed by one administration of saline solution one month apart.
  Interventions: Biological: Tetanus, reduced diphtheria, and acellular pertussis vaccine (adsorbed); Other: Saline solution
- Group 8: TdaP booster (Experimental): Subjects received tetanus, reduced diphtheria, and acellular pertussis vaccine (adsorbed) with different antigen dose formulations: medium dose of PT, FHA, PRN, double dose of D toxoid, fixed dose of T toxoid, followed by one administration of saline solution one month apart.
  Interventions: Biological: Tetanus, reduced diphtheria, and acellular pertussis vaccine (adsorbed); Other: Saline solution
- Group 9: TDaP booster (Experimental): Subjects received tetanus, reduced diphtheria, and acellular pertussis vaccine (adsorbed) with different antigen dose formulations: high dose of PT, FHA, PRN, double dose of D toxoid, fixed dose of T toxoid, followed by one administration of saline solution one month apart.
  Interventions: Biological: Tetanus, reduced diphtheria, and acellular pertussis vaccine (adsorbed); Other: Saline solution
- Group 10: Licensed TdaP booster (Active Comparator): Subject received one dose of a licensed TdaP booster vaccine (containing 8 μg each of PT, FHA and 2.5 μg of PRN antigens and 2.5 Lf of diphtheria toxoid and 5 Lf of tetanus toxoid) followed by one administration of saline solution one month apart.
  Interventions: Biological: Licensed TdaP booster vaccine; Other: Saline solution

INTERVENTIONS:
Biological: Acellular pertussis vaccine — Acellular pertussis (aP) vaccine was administered with different antigen doses intramuscularly in the upper deltoid region of the subject's non-dominant arm.
  Arms: Group 1: aP booster; Group 2: aP booster; Group 3: aP booster
Biological: Tetanus, reduced diphtheria, and acellular pertussis vaccine (adsorbed) — Tetanus, reduced diphtheria, and acellular pertussis (TdaP) vaccine was administered with different antigen doses intramuscularly in the upper deltoid region of the subject's non-dominant arm.
  Arms: Group 4: TdaP booster; Group 5: TdaP booster; Group 6: TdaP booster; Group 7: TdaP booster; Group 8: TdaP booster; Group 9: TDaP booster
Biological: Licensed TdaP booster vaccine — Licenced TdaP booster vaccine was administered intramuscularly in the upper deltoid region of the subject's non-dominant arm.
  Arms: Group 10: Licensed TdaP booster
Biological: Diphtheria and tetanus vaccine (adsorbed, reduced antigen content, Germany) — To ensure all subjects receive a tetanus and diphtheria booster vaccination, an injection was administered on Study Day 30, one month after the administration of the investigational vaccine.
  Arms: Group 1: aP booster; Group 2: aP booster; Group 3: aP booster
Other: Saline solution — Subjects received one injection of saline solution at one month after vaccination.
  Arms: Group 10: Licensed TdaP booster; Group 4: TdaP booster; Group 5: TdaP booster; Group 6: TdaP booster; Group 7: TdaP booster; Group 8: TdaP booster; Group 9: TDaP booster

SUMMARY:
This study will evaluate the safety and efficacy of 9 different vaccines containing aP (acellular pertussis) and TdaP (acellular pertussis, tetanus and diphtheria) in healthy subjects 18 to 40 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female individuals between 18 and 40 years of age (inclusive) who had provided informed consent.
2. Individuals who were able to be contacted for the duration of the study.

Exclusion Criteria:

1. Individuals who had received vaccines containing T, D, or pertussis (aP or whole cell), been diagnosed with pertussis disease, or who have had a household exposure to pertussis within the past 8 years.
2. If female, "of childbearing potential", sexually active, and had not used any of the "acceptable contraceptive methods" for at least 2 months prior to study entry:

   1. Of childbearing potential was defined as status post onset of menarche and not meeting any of the following conditions: menopausal for at least 2 years, status after bilateral tubal ligation for at least 1 year, status after bilateral oophorectomy, or status after hysterectomy.
   2. Acceptable birth control methods were defined as one or more of the following:

      * Hormonal contraceptive (such as oral, injection, transdermal patch, implant, cervical ring);
      * Barrier (condom with spermicide or diaphragm with spermicide) each and every time during intercourse;
      * Intrauterine device (IUD);
      * Monogamous relationship with vasectomized partner. Partner must have been vasectomized for at least six months prior to the subject's study entry.
3. If female of childbearing potential and sexually active, refusal to use an "acceptable contraceptive method" through to 3 weeks after last study vaccination.
4. Any positive or indeterminate pregnancy test.
5. Female individuals who were pregnant or breastfeeding.
6. Individuals with contraindications, warnings and/or precautions to vaccination with Boostrix or Td-pur as specified within the summary of product characteristics.
7. Individuals with a clinically significant active infection (as assessed by the investigator) or oral body temperature ≥38°C/100.4ºF within 3 days of the intended date of vaccination.
8. Known hypersensitivity or allergy to diphtheria, tetanus, or pertussis vaccine (including excipients of the investigational study vaccines, control or placebo as summarized in protocol section 5.0).
9. Individuals with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, might have interfered with the subject's ability to participate in the study.
10. Individuals with any progressive or severe neurologic disorder, seizure disorder or Guillian-Barré syndrome.
11. Individuals with history or any illness that, in the opinion of the investigator, might have interfered with the results of the study or pose additional risk to the individuals due to participation in the study.
12. Known or suspected impairment/alteration of immune function, including:

    1. Chronic use of oral steroids (≥15 days of use) within 60 days prior to visit 1 (day 1) (use of inhaled, intranasal, or topical corticosteroids was allowed);
    2. Receipt of parenteral steroids within 60 days prior to visit 1 (day 1);
    3. Receipt of immunostimulants within 60 days prior to visit 1 (day 1);
    4. Receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivates within 3 months prior to visit 1 (day 1) or planned during the full length of the study;
    5. HIV infection or HIV-related disease;
    6. Heritable immunodeficiency.
13. Abnormalities of splenic or thymic function.
14. Individuals with a known bleeding diathesis, or any condition that might have been associated with a prolonged bleeding time.
15. Individuals with any serious chronic or progressive disease according to judgment of the investigator (neoplasm, insulin dependent diabetes, cardiac, renal or hepatic disease).
16. Individuals with body mass index (BMI) greater than or equal to 35 kg/m2 (= weight in kg / (height in meters x height in meters)).
17. Individuals participating in any clinical trial with another investigational product 30 days prior to first study visit or with intent to participate in another clinical study at any time during the conduct of this study.
18. Individuals who received any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment in this study or who were planning to receive any vaccine other than Td or placebo within 28 days from the study vaccines.
19. Individuals who were first degree relatives of subjects involved in trial conduct.
20. Individuals with history of substance or alcohol abuse within the past 2 years.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 420 (Actual)
Dates: Start 2012-03; Primary Completion 2012-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines; Geert Leroux-Roels, Prof. Dr., Principal Investigator — Center for Vaccinology (CEVAC), Ghent University Hospital
Locations (1):
- Center for Vaccinology (CEVAC), Ghent University Hospital, De Pintelaan, B-9000 Ghent, Belgium

REFERENCES:
- [Derived] Leroux-Roels G, Lattanzi M, Solis CD, Contorni M, Costantini M, Moraschini L, Bardelli M, Bertholet S, Borgogni E, Buricchi F, Cantisani R, Faenzi E, Finco O, Leuzzi R, Pizza M, Rosa D, Schiavetti F, Seubert A, Spensieri F, Volpini G, Zedda L, Giudice GD, Galgani I. A phase I, randomized, controlled, dose-ranging study of investigational acellular pertussis (aP) and reduced tetanus-diphtheria-acellular pertussis (TdaP) booster vaccines in adults. Hum Vaccin Immunother. 2018 Jan 2;14(1):45-58. doi: 10.1080/21645515.2017.1385686. Epub 2017 Nov 27. PMID 29172945

RESULTS

PARTICIPANT FLOW:
Groups:
- Group aP1: Subjects received a single dose of aP booster vaccine (containing a low dose of PT, FHA and PRN antigens) on day 1 of this study.
- Group aP2: Subjects received a single dose of aP booster vaccine (containing a medium dose of PT, FHA and PRN antigens) on day 1 of this study.
- Group aP4: Subjects received a single dose of aP booster vaccine (containing a high dose of PT, FHA and PRN antigens) on day 1 of this study.
- Group T5D2aP1: Subjects received a single dose of TdaP booster vaccine (containing a low dose of PT, FHA, PRN antigens, a low dose of diphtheria toxoid a fixed dose of tetanus toxoid) on day 1 of this study.
- Group T5D2aP2: Subjects received a single dose of TdaP booster vaccine (containing a medium dose of PT, FHA, PRN antigens, a low dose of diphtheria toxoid and a fixed dose of tetanus toxoid) on day 1 of this study.
- Group T5D2aP4: Subjects received a single dose of TdaP booster vaccine (containing a high dose of PT, FHA, PRN antigens, a low dose of diphtheria toxoid and a fixed dose of tetanus toxoid) on day 1 of this study.
- Group T5D4aP1: Subjects received a single dose of TdaP booster vaccine (containing a low dose of PT, FHA, PRN antigens, a double dose of diphtheria toxoid and a fixed dose of tetanus toxoid) on day 1 of this study.
- Group T5D4aP2: Subjects received a single dose of TdaP booster vaccine (containing a medium dose of PT, FHA, PRN antigens, a double dose of diphtheria toxoid and a fixed dose of tetanus toxoid) on day 1 of this study.
- Group T5D4aP4: Subjects received a single dose of TdaP booster vaccine (containing a high dose of PT, FHA, PRN antigens, a double dose of diphtheria toxoid and a fixed dose of tetanus toxoid) on day 1 of this study.
- Licensed TdaP: Subjects received a single dose of a comparator TdaP booster vaccine (containing 8 μg each of PT, FHA and 2.5 μg of PRN antigens and 2.5 Lf of diphtheria toxoid and 5 Lf of tetanus toxoid) on day 1 of this study.
Period: Overall Study
Arm/Group | Group aP1 | Group aP2 | Group aP4 | Group T5D2aP1 | Group T5D2aP2 | Group T5D2aP4 | Group T5D4aP1 | Group T5D4aP2 | Group T5D4aP4 | Licensed TdaP
Started | 42 | 42 | 42 | 42 | 42 | 42 | 42 | 42 | 42 | 42
Completed | 40 | 41 | 40 | 40 | 40 | 41 | 40 | 42 | 41 | 42
Not Completed | 2 | 1 | 2 | 2 | 2 | 1 | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 1 | 0
Not completed — SAE - Premature contractions | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was done on the all enrolled set, ie, all subjects who have signed an informed consent, undergone screening procedures and were randomized.
Groups:
- Group T5D2aP1: Subjects received a single dose of TdaP booster vaccine (containing a low dose of PT, FHA, PRN antigens, a low dose of diphtheria toxoid and a fixed dose of tetanus toxoid) on day 1 of this study.
- Total: Total of all reporting groups
Arm/Group | Group aP1 | Group aP2 | Group aP4 | Group T5D2aP1 | Group T5D2aP2 | Group T5D2aP4 | Group T5D4aP1 | Group T5D4aP2 | Group T5D4aP4 | Licensed TdaP | Total
Number analyzed (Participants) | 42 | 42 | 42 | 42 | 42 | 42 | 42 | 42 | 42 | 42 | 420
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.6 (5.6) | 26.8 (5.1) | 27.4 (6.5) | 26.8 (5.7) | 27.7 (5.9) | 25.8 (5.2) | 25.1 (4.2) | 27.5 (5.1) | 27.2 (5.6) | 27.4 (6.4) | 26.8 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 28 | 25 | 23 | 27 | 24 | 29 | 19 | 27 | 24 | 250
  Male | 18 | 14 | 17 | 19 | 15 | 18 | 13 | 23 | 15 | 18 | 170

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects Reporting Solicited Local and Systemic Adverse Events After Receiving Different Formulations of aP and TdaP Booster Vaccine
Description: The safety profiles of different antigenic formulations of the aP and TdaP booster vaccines were assessed and compared to that of licensed comparator in terms of the number of subjects reporting solicited local and systemic adverse events and other adverse events after vaccination.
Time Frame: Day 1 through 7 after vaccination
Population: Analysis was done on the safety set, ie, all subjects who received the study vaccination and provided post vaccination safety data.
Measure: Number; unit: participants
Arm/Group | Group aP1 | Group aP2 | Group aP4 | Group T5D2aP1 | Group T5D2aP2 | Group T5D2aP4 | Group T5D4aP1 | Group T5D4aP2 | Group T5D4aP4 | Licensed TdaP
Number analyzed (Participants) | 42 | 42 | 41 | 42 | 42 | 42 | 41 | 42 | 42 | 42
participants
  Any local | 30 | 33 | 32 | 35 | 38 | 37 | 40 | 36 | 39 | 33
  Injection site erythema | 0 | 1 | 1 | 1 | 2 | 6 | 3 | 2 | 4 | 3
  Injection site induration | 3 | 3 | 1 | 6 | 1 | 7 | 9 | 4 | 4 | 6
  Injection site pruritus | 0 | 4 | 1 | 3 | 2 | 5 | 3 | 3 | 6 | 5
  Injection site pain | 30 | 32 | 31 | 35 | 38 | 36 | 40 | 35 | 39 | 31
  Any Systemic | 27 | 20 | 20 | 18 | 20 | 23 | 27 | 21 | 27 | 21
  Nausea | 3 | 6 | 2 | 1 | 2 | 5 | 4 | 6 | 7 | 1
  Fatigue | 19 | 14 | 13 | 13 | 15 | 18 | 20 | 15 | 16 | 12
  Generalized myalgia | 10 | 8 | 4 | 8 | 10 | 11 | 12 | 8 | 9 | 11
  Generalized arthralgia | 2 | 0 | 3 | 4 | 1 | 3 | 4 | 4 | 7 | 1
  Headache | 17 | 13 | 12 | 8 | 13 | 13 | 16 | 14 | 17 | 13
  Any Other | 6 | 7 | 2 | 6 | 8 | 4 | 8 | 7 | 7 | 8
  Body temperature (≥40°C) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Prophylactic use of analgesic/antipyretic | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 2 | 1
  Therapeutic use of analgesic/antipyretic | 6 | 7 | 2 | 6 | 8 | 3 | 8 | 7 | 7 | 8

2. Primary Outcome: The Number of Subjects Reporting Unsolicited Adverse Events After Receiving Different Formulations of aP and TdaP Booster Vaccine
Description: The safety profiles of different antigenic formulations of the aP and TdaP booster vaccines were assessed in terms of the number of subjects reporting any unsolicited adverse events (AEs) between day 1 to day 30 , serious adverse events (SAEs) and AEs leading to premature withdrawal between day 1 to day 365, after vaccination.
Time Frame: From day 1 to day 365
Population: Analysis was done on the safety set.
Measure: Number; unit: participants
Arm/Group | Group aP1 | Group aP2 | Group aP4 | Group T5D2aP1 | Group T5D2aP2 | Group T5D2aP4 | Group T5D4aP1 | Group T5D4aP2 | Group T5D4aP4 | Licensed TdaP
Number analyzed (Participants) | 42 | 42 | 41 | 42 | 42 | 42 | 41 | 42 | 42 | 42
participants
  Any AE (day 1 to 30) | 20 | 28 | 12 | 21 | 13 | 17 | 16 | 14 | 18 | 18
  At least possibly related unsolicited AEs | 11 | 13 | 7 | 8 | 9 | 11 | 7 | 4 | 11 | 10
  Any SAE (Day1 to Day 365) | 4 | 1 | 1 | 1 | 0 | 1 | 1 | 2 | 2 | 1
  At least possibly related SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AEs leading to withdrawal (Day1 to Day 365) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Geometric Mean Concentrations (GMCs) of Antibodies in aP1, aP2, aP4 Groups Against Pertussis Antigens Following Booster Vaccination
Description: The GMCs of antibodies as measured by enzyme-linked immunosorbent assay (ELISA) on aP booster groups, against pertussis antigens pertussis toxoid (PT), filamentous hemagglutinin (FHA), pertactin (PRN), following vaccination with different antigenic formulations of aP versus the response to the commercially available comparator are reported.
Time Frame: Day 1 (baseline) and Day 30 post vaccination
Population: Analysis was done on the per-protocol population, ie, all subjects who correctly received the vaccine, and provided evaluable serum samples at the relevant time points and had no major protocol violation as defined prior to unblinding.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Groups:
- Licensed TdaP: Subjects received a single dose of a comparator TdaP booster vaccine (containing 8 μg each of PT, FHA and 2.5 μg of PRN antigens and 2.5 Lf of diphtheria toxoid and 5 Lf of tetanus toxoid) on day1 of this study.
Arm/Group | Group aP1 | Group aP2 | Group aP4 | Licensed TdaP
Number analyzed (Participants) | 42 | 38 | 39 | 40
µg/mL
  Day 1 (PT) | 4.92 [3.22 to 7.53] | 3.81 [2.43 to 5.95] | 4.23 [2.72 to 6.57] | 5.07 [3.28 to 7.84]
  Day 30 (PT; N= 39,35,36,40) | 91 [67 to 122] | 145 [106 to 199] | 182 [133 to 249] | 87 [65 to 117]
  Day 1 (FHA) | 20 [15 to 27] | 16 [11 to 22] | 21 [15 to 29] | 20 [15 to 28]
  Day 30 (FHA; N= 39,35,36,40) | 114 [93 to 140] | 147 [119 to 182] | 183 [148 to 226] | 241 [198 to 294]
  Day 1 (PRN) | 20 [14 to 28] | 16 [11 to 23] | 17 [12 to 25] | 21 [14 to 31]
  Day 30 (PRN; N= 39,35,36,40) | 589 [440 to 788] | 936 [687 to 1273] | 1384 [1020 to 1878] | 475 [356 to 635]

4. Primary Outcome: GMCs of Antibodies in T5D2aP1, T5D2aP2 and T5D2aP4 Groups Against Pertussis Antigens Following Booster Vaccination
Description: The GMCs of antibodies as measured by enzyme-linked immunosorbent assay (ELISA) in TdaP Booster Groups against pertussis antigens (PT, FHA and PRN), following vaccination with different antigenic formulations of TdaP booster versus the response to the commercially available comparator are reported.
Time Frame: Day 1 (baseline) and Day 30 post vaccination
Population: Analysis was done on the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Group T5D2aP1 | Group T5D2aP2 | Group T5D2aP4 | Licensed TdaP
Number analyzed (Participants) | 41 | 38 | 40 | 40
µg/mL
  Day 1 (PT) | 4.35 [2.86 to 6.6] | 4.97 [3.22 to 7.67] | 4.8 [3.15 to 7.32] | 5.07 [3.32 to 7.73]
  Day 30 (PT; N= 41,38,38,40) | 62 [49 to 80] | 72 [56 to 93] | 160 [124 to 206] | 86 [68 to 110]
  Day 1 (FHA) | 20 [14 to 28] | 16 [12 to 23] | 23 [17 to 33] | 20 [15 to 28]
  Day 30 (FHA; N= 41,38,38,40) | 83 [69 to 100] | 90 [74 to 109] | 118 [97 to 143] | 241 [200 to 291]
  Day 1 (PRN) | 13 [8.72 to 21] | 21 [13 to 32] | 27 [17 to 41] | 21 [14 to 32]
  Day 30 (PRN; N= 41,38,38,40) | 445 [317 to 626] | 803 [567 to 1138] | 1092 [766 to 1555] | 496 [353 to 696]

5. Primary Outcome: GMCs of Antibodies in T5D4aP1, T5D4aP2 and T5D4aP4 Groups Against Pertussis Antigens Following Vaccination
Description: The GMCs of antibodies as measured by enzyme-linked immunosorbent assay (ELISA) in TdaP booster groups, against pertussis antigens (PT, FHA and PRN), following vaccination with different antigenic formulations of TdaP booster versus the response to the commercially available comparator are reported.
Time Frame: Day 1 (baseline) and Day 30 post vaccination
Population: Analysis was done on the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Group T5D4aP1 | Group T5D4aP2 | Group T5D4aP4 | Licensed TdaP
Number analyzed (Participants) | 37 | 39 | 40 | 40
µg/mL
  Day 1 (PT) | 8.74 [5.64 to 14] | 8.2 [5.32 to 13] | 8.06 [5.25 to 12] | 5.07 [3.3 to 7.78]
  Day 30 (PT) | 83 [64 to 108] | 93 [72 to 120] | 157 [122 to 202] | 93 [72 to 119]
  Day 1 (FHA) | 24 [17 to 33] | 27 [20 to 38] | 26 [18 to 36] | 20 [15 to 28]
  Day 30 (FHA) | 116 [96 to 140] | 100 [83 to 121] | 113 [94 to 135] | 252 [210 to 303]
  Day 1 (PRN) | 30 [20 to 47] | 22 [14 to 34] | 28 [19 to 43] | 21 [14 to 32]
  Day 30 (PRN) | 837 [624 to 1124] | 680 [510 to 906] | 1024 [772 to 1359] | 506 [381 to 671]

6. Secondary Outcome: Percentages of Subjects With 2- and 4-fold Increase in GMCs Against Pertussis Antigens Following Vaccination.
Description: Comparison of antibody responses against pertussis antigens (PT, FHA and PRN), following vaccination with different antigenic formulations of aP and TdaP booster vaccines and licensed comparator, are reported in terms of the percentages of subjects demonstrating 2- and 4-fold increase in GMCs from baseline.
Time Frame: Day 30 post vaccination
Population: Analysis was done on the per-protocol population.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group aP1 | Group aP2 | Group aP4 | Group T5D2aP1 | Group T5D2aP2 | Group T5D2aP4 | Group T5D4aP1 | Group T5D4aP2 | Group T5D4aP4 | Licensed TdaP
Number analyzed (Participants) | 39 | 35 | 36 | 41 | 38 | 38 | 37 | 39 | 40 | 40
percentage of subjects
  2-Fold (PT) | 100 [91 to 100] | 100 [90 to 100] | 94 [81 to 99] | 95 [83 to 99] | 95 [82 to 99] | 100 [91 to 100] | 89 [75 to 97] | 90 [76 to 97] | 95 [83 to 99] | 100 [91 to 100]
  4-Fold (PT) | 92 [79 to 98] | 100 [90 to 100] | 92 [78 to 98] | 80 [65 to 91] | 76 [60 to 89] | 100 [91 to 100] | 81 [65 to 92] | 77 [61 to 89] | 93 [80 to 98] | 98 [87 to 100]
  2-Fold (FHA) | 85 [69 to 94] | 94 [81 to 99] | 89 [74 to 97] | 80 [65 to 91] | 95 [82 to 99] | 95 [82 to 99] | 76 [59 to 88] | 77 [61 to 89] | 90 [76 to 97] | 95 [83 to 99]
  4-Fold (FHA) | 59 [42 to 74] | 83 [66 to 93] | 83 [67 to 94] | 46 [31 to 63] | 61 [43 to 76] | 58 [41 to 74] | 46 [29 to 63] | 56 [40 to 72] | 53 [36 to 68] | 83 [67 to 93]
  2-Fold (PRN) | 100 [91 to 100] | 100 [90 to 100] | 100 [90 to 100] | 98 [87 to 100] | 100 [91 to 100] | 100 [91 to 100] | 97 [86 to 100] | 92 [79 to 98] | 100 [91 to 100] | 100 [91 to 100]
  4-Fold (PRN) | 92 [79 to 98] | 100 [90 to 100] | 100 [90 to 100] | 90 [77 to 97] | 95 [82 to 99] | 97 [86 to 100] | 89 [75 to 97] | 85 [69 to 94] | 98 [87 to 100] | 90 [76 to 97]

7. Secondary Outcome: GMCs of Antibodies Against Diphtheria and Tetanus Antigens Following Vaccination
Description: The GMCs of antibodies against diphtheria and tetanus antigens following vaccination with different formulations of TdaP booster are compared with the response to the commercially available comparator.
Time Frame: Day 1 (baseline) and Day 30 post vaccination
Population: Analysis was done on the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Group aP1 | Group aP2 | Group aP4 | Group T5D2aP1 | Group T5D2aP2 | Group T5D2aP4 | Group T5D4aP1 | Group T5D4aP2 | Group T5D4aP4 | Licensed TdaP
Number analyzed (Participants) | 39 | 35 | 36 | 41 | 38 | 38 | 37 | 39 | 40 | 40
IU/mL
  Day 1 (diphteria; N=42,38,39,41,38,40,37,39,40,40) | 0.4 [0.27 to 0.6] | 0.43 [0.28 to 0.65] | 0.25 [0.17 to 0.38] | 0.31 [0.2 to 0.46] | 0.15 [0.098 to 0.23] | 0.29 [0.19 to 0.44] | 0.31 [0.2 to 0.48] | 0.25 [0.16 to 0.39] | 0.25 [0.17 to 0.39] | 0.3 [0.19 to 0.45]
  Day 30 (diphteria) | 0.39 [0.32 to 0.49] | 0.39 [0.31 to 0.5] | 0.37 [0.29 to 0.46] | 1.48 [1.1 to 1.99] | 1.41 [1.04 to 1.92] | 1.63 [1.2 to 2.21] | 2.7 [1.97 to 3.69] | 2.19 [1.62 to 2.97] | 2.47 [1.83 to 3.33] | 1.79 [1.32 to 2.41]
  Day 1 (tetanus; N=42,38,39,41,38,40,37,39,40,40) | 2.45 [1.9 to 3.16] | 2.11 [1.61 to 2.76] | 2.27 [1.74 to 2.96] | 1.93 [1.44 to 2.58] | 1.99 [1.47 to 2.68] | 2.07 [1.54 to 2.77] | 2.04 [1.5 to 2.76] | 2.62 [1.95 to 3.53] | 1.92 [1.43 to 2.58] | 1.89 [1.41 to 2.53]
  Day 30 (tetanus) | 2.19 [1.91 to 2.52] | 2.18 [1.88 to 2.52] | 2.19 [1.89 to 2.53] | 8.15 [6.73 to 9.88] | 8.82 [7.23 to 11] | 7.01 [5.74 to 8.56] | 8.23 [6.73 to 10] | 6.82 [5.6 to 8.32] | 7.44 [6.13 to 9.04] | 8.49 [6.99 to 10]

8. Secondary Outcome: GMRs of Post Vaccination Versus Pre Vaccination GMCs of Antibodies Against Diphtheria and Tetanus Antigens
Description: The GMRs of post vaccination versus pre vaccination GMCs of antibodies against diphtheria and tetanus antigens for different formulations of TdaP booster and commercially available comparator versus GMCs at baseline are reported.
Time Frame: Day 30 post vaccination/Day 1
Population: Analysis was done on the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Group aP1 | Group aP2 | Group aP4 | Group T5D2aP1 | Group T5D2aP2 | Group T5D2aP4 | Group T5D4aP1 | Group T5D4aP2 | Group T5D4aP4 | Licensed TdaP
Number analyzed (Participants) | 39 | 35 | 36 | 41 | 38 | 38 | 37 | 39 | 40 | 40
Ratio
  Day 30/day 1 (diphtheria) | 1.05 [0.94 to 1.16] | 1.05 [0.93 to 1.17] | 1.19 [1.07 to 1.33] | 5.24 [3.66 to 7.49] | 8.58 [5.91 to 12] | 5.62 [3.87 to 8.16] | 9.18 [6.3 to 13] | 8.39 [5.81 to 12] | 9.54 [6.64 to 14] | 6.1 [4.25 to 8.78]
  Day 30/day 1 (tetanus) | 0.94 [0.88 to 1.02] | 0.92 [0.86 to 1] | 0.97 [0.9 to 1.04] | 4.2 [3.01 to 5.86] | 4.43 [3.14 to 6.26] | 3.43 [2.43 to 4.84] | 4.02 [2.83 to 5.71] | 2.64 [1.88 to 3.71] | 3.86 [2.76 to 5.41] | 4.5 [3.21 to 6.3]

9. Primary Outcome: Geometric Mean Ratios (GMRs) of Post Vaccination Versus Pre Vaccination GMCs of Antibodies in aP1, aP2, aP4 Booster Groups Against Pertussis Antigens
Description: The GMRs of post-vaccination versus pre-vaccination GMCs of antibodies against pertussis antigens (PT, FHA and PRN) for different antigenic formulations of aP booster vaccines and for licensed comparator are reported.
Time Frame: Day 30 post vaccination/baseline (Day 1)
Population: Analysis was done on the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Group aP1 | Group aP2 | Group aP4 | Licensed TdaP
Number analyzed (Participants) | 39 | 35 | 36 | 40
Ratio
  Day 30/Day 1 (PT) | 18 [12 to 26] | 36 [24 to 54] | 49 [33 to 73] | 17 [12 to 25]
  Day 30/Day 1 (FHA) | 5.49 [3.99 to 7.54] | 9.42 [6.74 to 13] | 9.39 [6.75 to 13] | 12 [8.73 to 16]
  Day 30/Day 1 (PRN) | 30 [21 to 44] | 58 [39 to 86] | 81 [54 to 119] | 24 [16 to 34]

10. Primary Outcome: GMRs of Post Vaccination Versus Pre Vaccination GMCs of Antibodies in T5D2aP1, T5D2aP2 and T5D2aP4 Booster Groups Against Pertussis Antigens
Description: The GMRs of post-vaccination versus pre-vaccination GMCs of antibodies against pertussis antigens (PT, FHA and PRN) for TdaP booster groups and for licensed comparator are reported.
Time Frame: Day 30 post vaccination/baseline (Day 1)
Population: Analysis was done on the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Group T5D2aP1 | Group T5D2aP2 | Group T5D2aP4 | Licensed TdaP
Number analyzed (Participants) | 41 | 38 | 38 | 40
Ratio
  Day 30/Day 1 (PT) | 14 [9.58 to 21] | 15 [10 to 23] | 31 [21 to 46] | 17 [12 to 26]
  Day 30/Day 1 (FHA) | 4.24 [3.21 to 5.6] | 5.02 [3.76 to 6.71] | 5.11 [3.83 to 6.83] | 12 [9.01 to 16]
  Day 30/Day 1 (PRN) | 30 [21 to 45] | 38 [25 to 57] | 46 [31 to 69] | 24 [16 to 35]

11. Primary Outcome: GMRs of Post Vaccination Versus Pre Vaccination GMCs of Antibodies for T5D4aP1, T5D4aP2 and T5D4aP4 Booster Groups Against Pertussis Antigens
Description: as for outcome 10
Time Frame: Day 30 post vaccination/baseline (Day 1)
Population: Analysis was done on the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Group T5D4aP1 | Group T5D4aP2 | Group T5D4aP4 | Licensed TdaP
Number analyzed (Participants) | 37 | 39 | 40 | 40
Ratio
  Day 30/Day 1 (PT) | 9.51 [6.38 to 14] | 12 [7.9 to 17] | 20 [14 to 29] | 17 [12 to 25]
  Day 30/Day 1 (FHA) | 4.7 [3.47 to 6.38] | 3.95 [2.94 to 5.31] | 4.39 [3.28 to 5.89] | 12 [8.91 to 16]
  Day 30/Day 1 (PRN) | 27 [18 to 42] | 32 [21 to 48] | 36 [24 to 54] | 24 [16 to 36]

12. Primary Outcome: Percentages of Subjects With Diphtheria and Tetanus Antitoxin Units >= 0.1/mL After Vaccination
Description: The percentages of subjects demonstrating diphtheria and tetanus antitoxin units >= 0.1/mL following vaccination with different antigenic formulations of TdaP booster vaccine, is compared to the response to commercially available comparator.
Time Frame: Day 1 (baseline) and Day 30 post vaccination
Population: Analysis was done on the per-protocol population.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | Group aP1 | Group aP2 | Group aP4 | Group T5D2aP1 | Group T5D2aP2 | Group T5D2aP4 | Group T5D4aP1 | Group T5D4aP2 | Group T5D4aP4 | Licensed TdaP
Number analyzed (Participants) | 39 | 35 | 36 | 41 | 38 | 38 | 37 | 39 | 40 | 40
percentages of subjects
  Day 1 (diphteria; N=42,38,39,41,38,40,37,39,40,40) | 79 [63 to 90] | 89 [75 to 97] | 72 [55 to 85] | 71 [54 to 84] | 68 [51 to 82] | 85 [70 to 94] | 81 [65 to 92] | 72 [55 to 85] | 78 [62 to 89] | 80 [64 to 91]
  Day 30 (diphteria) | 87 [73 to 96] | 97 [85 to 100] | 81 [64 to 92] | 98 [87 to 100] | 97 [86 to 100] | 95 [82 to 99] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100]
  Day 1 (tetanus; N=42,38,39,41,38,40,37,39,40,40) | 98 [87 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 95 [83 to 99] | 100 [91 to 100] | 100 [91 to 100] | 98 [87 to 100] | 95 [83 to 99]
  Day 30 (tetanus) | 100 [91 to 100] | 100 [90 to 100] | 100 [90 to 100] | 100 [91 to 100] | 100 [91 to 100] | 97 [86 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100] | 100 [91 to 100]

ADVERSE EVENTS:
Time Frame: Solicited and unsolicited AEs collected from Day 1 to Day 7; SAEs, medically attended AEs and AEs leading to withdrawal collected from Day 1 to Day 365.
Description: Analysis was done on the safety population; two subjects, in groups aP4 and T5D4aP1were excluded for not providing any postbaseline safety data. Solicited AEs are categorized as systematic and unsolicited AEs are categorized as non-systematic.
Arm/Group | Group aP1 | Group aP2 | Group aP4 | Group T5D2aP1 | Group T5D2aP2 | Group T5D2aP4 | Group T5D4aP1 | Group T5D4aP2 | Group T5D4aP4 | Licensed TdaP
Serious Adverse Events (participants affected / at risk) | 4/42 | 1/42 | 1/41 | 1/42 | 0/42 | 1/42 | 1/41 | 2/42 | 2/42 | 1/42
Other Adverse Events (participants affected / at risk) | 36/42 | 39/42 | 36/41 | 38/42 | 41/42 | 42/42 | 40/41 | 39/42 | 40/42 | 36/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group aP1 (N=42) | Group aP2 (N=42) | Group aP4 (N=41) | Group T5D2aP1 (N=42) | Group T5D2aP2 (N=42) | Group T5D2aP4 (N=42) | Group T5D4aP1 (N=41) | Group T5D4aP2 (N=42) | Group T5D4aP4 (N=42) | Licensed TdaP (N=42)
Peritonsillar abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysthymic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group aP1 (N=42) | Group aP2 (N=42) | Group aP4 (N=41) | Group T5D2aP1 (N=42) | Group T5D2aP2 (N=42) | Group T5D2aP4 (N=42) | Group T5D4aP1 (N=41) | Group T5D4aP2 (N=42) | Group T5D4aP4 (N=42) | Licensed TdaP (N=42)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 1 | 3 | 0 | 2 | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 6 | 2 | 2 | 2 | 5 | 4 | 6 | 7 | 1
Axillary pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 19 | 14 | 13 | 13 | 15 | 18 | 21 | 15 | 16 | 12
Injection site erythema (General disorders) | 0 | 2 | 1 | 1 | 1 | 7 | 2 | 1 | 4 | 3
Injection site induration (General disorders) | 2 | 4 | 1 | 3 | 1 | 6 | 8 | 4 | 3 | 5
Injection site movement impairment (General disorders) | 2 | 3 | 2 | 2 | 2 | 1 | 3 | 2 | 0 | 1
Injection site pain (General disorders) | 30 | 32 | 31 | 35 | 38 | 36 | 40 | 35 | 39 | 31
Injection site pruritus (General disorders) | 0 | 4 | 1 | 3 | 2 | 5 | 3 | 3 | 6 | 5
Pyrexia (General disorders) | 1 | 0 | 2 | 2 | 1 | 1 | 3 | 2 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 5 | 5 | 2 | 4 | 1 | 3 | 3 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 4 | 1 | 3 | 5 | 4 | 8 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 9 | 4 | 8 | 10 | 12 | 14 | 8 | 9 | 11
Headache (Nervous system disorders) | 19 | 15 | 13 | 9 | 14 | 13 | 16 | 15 | 19 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 4 | 0 | 2 | 3 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days